CLINICAL TRIAL: NCT02570737
Title: Latin American Pulmonary Hypertension Registry
Acronym: RELAHP
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Asociacion Latinoamericana de Torax (Industry)
Collaborators: Actelion (Industry); Bayer (Industry); Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: Cardioneumology
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Incident patients: Patients with less than three months from diagnosis to start of the Registry or those who have been diagnosed during the recruitment period.
- Prevalent patients: Patients who have been diagnosed with more than three months from diagnosis to start of the Registry.

SUMMARY:
The RELAHP registry is a Latin-American multinational, multicenter, prospective observational registry-type cohort study, which pretends to identify clinical characteristics, clinical course, management and outcome of all forms of pulmonary hypertension (PH).

All consecutively consented patients newly diagnosed with WHO Group I-V PH according to specific hemodynamic criteria on right heart catheterization at the participating centers will be enrolled. Patients will be followed six-monthly for a minimum of five years from the time of enrollment.

DETAILED DESCRIPTION:
Introduction. Pulmonary hypertension (PH) is a worldwide group of vascular diseases characterized by progressive increase in pulmonary vascular resistance and pulmonary arterial pressure with secondary vascular and right ventricular (RV) remodeling, RV dysfunction, heart failure syndromes and, finally, premature death. In developed countries significant medical advances have occurred in the last two decades including a more systematic assessment and availability of new therapeutic approaches. In addition, current registries had shown new data regarding epidemiology, demography, clinical presentation, treatment and prognosis. However, the evidence coming from developing countries is scarce and more information is necessary to identify current care in such populations. In the other hand, high quality clinical registries may help to understand if the knowledge coming from clinical trials is being properly applied and if their results are reproducible in day-to-day clinical practice. The results of the REMEHIP, a registry with one-year enrollment and four-year follow-up will hopefully broad the investigators knowledge about clinical profile, medical care, therapeutic trends and outcome in a Mexican population with well characterized PH. Data collection will not only set current practices in relation to the epidemiology, diagnostics and treatment of PH in Latin-American, but will also set the mark for future investigations.

RELAHP itself is property of the Department of Pulmonary Circulation at the Latin American Thoracic Association (ALAT) and the participating doctors are members of this department. The registry is sponsored by ALAT with additional funding from multiple sponsors (Bayer Health Care, Actelion/Biotoscana, Grupo Ferrer).

RELAHP´s main objective is to shed light on the epidemiologic characteristics and clinical presentation of patients presenting with PH in Latin America, thus helping to know population evolution, all this by gathering the information, collected by main centers that work with PH in the region, on a uniform database. The data will allow establishing proper strategies for an early detection of the disease and a rational, therapeutic approach. Patients with newly diagnosed PH confirmed by right heart catheterization will be eligible for inclusion in the registry. This registry does not provide a predetermined appointment system; instead, the patient's treating doctor - according to the patients needs - shall determine the frequency of visits. Nevertheless, the record of condition and patient evolution must be actualized every six months.

Variables to be included. In all patients: a) date of onset of symptoms, b) medical history, c) treatment at enrollment, d) physical examination, d) WHO function class, e) six-minute walk distance, f) ECG, g) chest x-ray, h) echocardiogram, i) pulmonary function tests, j) V/Q lung scan and or pulmonary angiography, and/or pulmonary angiotomography k) right heart catheterization, and whenever possible indicated acute vasodilator challenge l) Laboratory test o) in-hospital and follow - up outcome, p) MACE q)Diagnostic classification l)Treatment intervention m)drug therapy, n)surgical interventions.

Visit office. Data will be collected in the first outcome and update through each follow-up about expected PH symptoms, functional class (WHO), current treatment, dose, compliance, collateral effects and concomitant medication, weight, blood pressure, heart and respiratory rate, and biomarkers, will be recorded in each visit.

Visits will be according with the standard health care of each center, but in general they will be made at least one every six months.

Quality Criteria. Following criteria will be used to improve quality data: a) standardized definitions, data and reports; b) tools for fast feedback; c) meetings among principal investigators and steering committee, at least one per year; d) ethics procedures review; e) electronic, simple and accessible data collection; f) rigorous center selection based on investigators expertise and/or facilities resources); g) consecutive patients enrollment to obtain representative sample; h) random centers audit; i) centralized data and statistical analysis; j) report all data and consistent conclusion; and k) transparency of funds for any publication. Furthermore, the quality of this registry will also be measured by the number of publications and presentations in national and international meetings as has previously been done.

Statistics. Quantitative baseline and continuous variables will be expressed as percentages, mean, standard deviation, odds ratio and CI. Differences between two groups will be examined by Student's t test and for multiple comparisons analysis of variance or nonparametric test. To analyze variables X2 will be used by Fisher's test. Cox proportional risk multivariate model will assess the relationship between each of these variables.

Structure of RELAHP: Executive committee, Single Data Centers (PH centers), Data Control Group and Publishing Group.

RELAHP is a multicenter project with doctors being the sole owners of the data of each individual PH center, and only the consolidated results, which are anonymous, are property of ALAT, thus keeping patient confidentiality and privacy safe.

As of 2014, a total of 12 centers (to be expanded) will contribute data to the registry during the planned five-year study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old
* Patients with any Group of Pulmonary Hypertension according to OMS Clinical Clasification (PH by RHC)
* Informed consent

Exclusion Criteria:

* Severe pulmonary function abnormalities (vital capacity < 60% predicted, FEV1 < 50% predicted)
* Abnormal pulmonary capillary wedge pressure (> 15 mmHg)
* Refusal to participate.
* Patients younger than 18 years old

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Latin American Patients of any age, with diagnosis of Pulmonary Hypertension from groups I-V confirmed by Right Heart Catheterization
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-07 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 5 years (Patients will be followed six-monthly for a minimum of five years)
  n-hospital or outpatient heart failure, cardiogenic shock, syncope, cardiovascular death and bleeding complications.

SECONDARY OUTCOMES:
Cardiovascular death | 5 years
  Secondary to right heart failure, cardiogenic shock, auricular or ventricular arrhythmia.

CONTACTS AND LOCATIONS:
Overall Officials: TOMAS R. PULIDO, M.D., Principal Investigator — ASOCIACIÓN LATINOAMERICANA DE TORAX
Locations (8):
- Hospital Universitario, Fundación Favaloro, Buenos Aires, Argentina
- Hospital Clementino Fraga - Universidade Federal do Rio de Janeiro, Rio de Janeiro, Brazil
- Instituto Nacional del Tórax, Universidad de Chile, Santiago, Chile
- Clínica Cardio Vid, Medellín, Colombia
- Honduras Medical Center, Tegucigalpa, Honduras
- Instituto Nacional de Cardiologia "Dr. Ignacio Chavez", Mexico City, Tlalpan, Mexico
- Hospital Maciel, Montevideo, Uruguay
- Hospital de Clínicas Caracas, Caracas, Venezuela

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Pulmonary Hypertension — https://www.nlm.nih.gov/medlineplus/pulmonaryhypertension.html
- See also: High Blood Pressure — https://www.nlm.nih.gov/medlineplus/highbloodpressure.html